CLINICAL TRIAL: NCT03413189
Title: PREDICTABLE: The Effect of Exercise Dosage on Physical Function, Cognition and Disability Following Critical Illness
Brief Title: The Effect of Exercise Dosage on Physical Function, Cognition and Disability Following Critical Illness
Acronym: PREDICTABLE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: Monash Health (Other); Monash University (Other)
Responsible Party: Sponsor
Other Study IDs: ANZICRC/PREDICTABLE/001
Record Dates: First submitted 2017-11-12; First posted 2018-01-29 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Critical Illness
Keywords: Exercise; Dosage; Function
MeSH Terms: conditions — Critical Illness; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PREDICT participants: This cohort is obtained from the PREDICT study enrolment (approx. 500) and a review of their medical records will be conducted
  Interventions: Other: Review of medical records
- PREDITCABLE participants: This is a nested cohort of patients recruited into PREDICT (approx. 40) that consent for a physiotherapist home visit to assess their physical and cognitive function and perform and interview to obtain themes regarding recovery
  Interventions: Other: Review of medical records; Other: Assessment of physical and cognitive function; Other: Interview of patients, carers and/or family members

INTERVENTIONS:
Other: Review of medical records — Medical records of patients will be reviewed to establish the median and highest level of functional achieved in Intensive Care (intensity) and the percentage of exercise sessions performed (frequency)
Other: Assessment of physical and cognitive function — This will be performed in person through the Function Independence Measure (FIM), grip strength, functional reach, 6-minute walk test (6MWT) and Montreal Cognitive Assessment (MoCA-Blind).
  Groups: PREDITCABLE participants
Other: Interview of patients, carers and/or family members — Questions will be asked to participants regarding their recovery from Intensive Care to establish themes
  Groups: PREDITCABLE participants

SUMMARY:
Survival following a critical illness continues to improve with ongoing developments in medical management, however evidence shows that this patient group is at a high risk of suffering long term disability. The objectives are to determine if there is a link between the amount of exercise performed in intensive care on the presence of delirium, long term cognition and disability whilst ensuring that patient reported outcomes correlate with actual measured results, and to obtain information on recovery from patients and/or relatives to determine themes.

DETAILED DESCRIPTION:
Survival from a critical illness is increasing, however the long term effect on patient's quality of life and the ability for patients to return to pre-illness function is unfavourable. Exercise in the ICU has been proven to be safe and effective, with decreases in length of stay and improvements in physical and psychosocial function seen in multiple studies. At present, the investigators are unsure on the most effective way to exercise this patient group in relation to duration, type, intensity and frequency.

The investigators aim to link the presence of delirium during an ICU admission, disability-free survival and quality of life obtained from telephone follow-up six months following ICU discharge with the amount of exercise performed during their ICU stay to determine a relationship. Additionally, in a small group of participants, the investigators will measure cognitive and physical function to ensure that the patient reported data accurately reflects their true functional level, while allowing patients and/or relatives, next of kin or carers to provide information regarding their recovery through an interview process.

The measure of physical function and disability (via the WHODAS and Euro Qol Group Health Survey (EQ5D)) obtained during telephone interview of the 500 patients enrolled in the PREDICT study will be correlated with the amount of exercise they performed whilst in Intensive Care obtained from the medical records. The presence of delirium will also be obtained from the medical records and linked with the amount of exercise performed to determine if a link is present. A sub-set of this population (40) will be invited at the 3-month follow up phone call of the PREDICT study to have a physiotherapist visit them to assess their cognitive and physical function and interview them and/or their relatives, next of kin or carer to determine themes of the recovery process following critical illness.

ELIGIBILITY:
Inclusion Criteria:

- ICU patients who have been invasively mechanically ventilated for over 24 hours

Exclusion Criteria:

* Patients aged less than 18 years old
* A proven or suspected acute primary brain process that is likely to result in global impairment of conscious level or cognition (e.g. Traumatic Brain Injury, Subarachnoid Haemorrhage, stroke or hypoxic brain injury after cardiac arrest)
* Second or subsequent admission to ICU during a single hospital admission
* Death is deemed imminent and inevitable
* Participants who do no not speak English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients who were mechanically ventilated > 24 hours in an intensive care unit who have survived to hospital discharge.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-03-09 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The measure the effect of exercise dosage in critical care on physical function | 6 months after ICU admission
  To correlate the amount of exercise performed in ICU on objectively measured physical function at 6 months following ICU admission (via 6MWT and FIM).
The measure the effect of exercise dosage in critical care on cognitive function | Up to 6 months following ICU admission
  To correlate the amount of exercise performed in ICU on cognitive function (via MoCA Blind)

SECONDARY OUTCOMES:
To correlate patient reported functional outcomes EQ5D with objectively measured outcomes | 6 months after ICU admission
  Compare patient reported disability score (EQ-5D) with a gold standard functional outcome measure (6MWT and FIM)
To correlate patient reported functional outcomes WHODAS with objectively measured outcomes | 6 months after ICU admission
  Compare patient reported disability score (WHODAS) with a gold standard functional outcome measure (6MWT and FIM).
Identify themes regarding recovery from critical illness from patient interviews | 6 months after ICU admission
  Compare qualitative data from patients and relatives/carers/next of kin to identify themes regarding the recovery process.
To correlate patient reported cognitive outcomes with in person measured cognitive outcomes | 6 months after ICU admission
  Compare patient reported MoCA Blind scores with those of the same test measured in person

CONTACTS AND LOCATIONS:
Overall Officials: Carol Hodgson, A/Prof, Principal Investigator — Australian and New Zealand intensive Care Reserch Centre
Locations (3):
- Australia (3):
  - Monash Medical Centre, Clayton, Victoria
  - Dandenong Hospital, Dandenong, Victoria
  - Australian and New Zealand Intensive Care Research Centre, Melbourne, Victoria

REFERENCES:
- [Background] Ali NA, O'Brien JM Jr, Hoffmann SP, Phillips G, Garland A, Finley JC, Almoosa K, Hejal R, Wolf KM, Lemeshow S, Connors AF Jr, Marsh CB; Midwest Critical Care Consortium. Acquired weakness, handgrip strength, and mortality in critically ill patients. Am J Respir Crit Care Med. 2008 Aug 1;178(3):261-8. doi: 10.1164/rccm.200712-1829OC. Epub 2008 May 29. PMID 18511703
- [Background] Angus DC, Musthafa AA, Clermont G, Griffin MF, Linde-Zwirble WT, Dremsizov TT, Pinsky MR. Quality-adjusted survival in the first year after the acute respiratory distress syndrome. Am J Respir Crit Care Med. 2001 May;163(6):1389-94. doi: 10.1164/ajrccm.163.6.2005123. PMID 11371406
- [Background] Thomas HC, Scully LJ, Lever AM, Yap I, Pignatelli M. A review of the efficacy of adenine arabinoside and lymphoblastoid interferon in the Royal Free Hospital studies of hepatitis B virus carrier treatment: identification of factors influencing response rates. Infection. 1987;15 Suppl 1:S26-31. doi: 10.1007/BF01650108. PMID 2439462
- [Background] Barnato AE, Albert SM, Angus DC, Lave JR, Degenholtz HB. Disability among elderly survivors of mechanical ventilation. Am J Respir Crit Care Med. 2011 Apr 15;183(8):1037-42. doi: 10.1164/rccm.201002-0301OC. Epub 2010 Nov 5. PMID 21057004
- [Background] Berney SC, Harrold M, Webb SA, Seppelt I, Patman S, Thomas PJ, Denehy L. Intensive care unit mobility practices in Australia and New Zealand: a point prevalence study. Crit Care Resusc. 2013 Dec;15(4):260-5. PMID 24289506
- [Background] Cheung AM, Tansey CM, Tomlinson G, Diaz-Granados N, Matte A, Barr A, Mehta S, Mazer CD, Guest CB, Stewart TE, Al-Saidi F, Cooper AB, Cook D, Slutsky AS, Herridge MS. Two-year outcomes, health care use, and costs of survivors of acute respiratory distress syndrome. Am J Respir Crit Care Med. 2006 Sep 1;174(5):538-44. doi: 10.1164/rccm.200505-693OC. Epub 2006 Jun 8. PMID 16763220
- [Background] Cuthbertson BH, Elders A, Hall S, Taylor J, MacLennan G, Mackirdy F, Mackenzie SJ; Scottish Critical Care Trials Group; Scottish Intensive Care Society Audit Group. Mortality and quality of life in the five years after severe sepsis. Crit Care. 2013 Apr 16;17(2):R70. doi: 10.1186/cc12616. PMID 23587132
- [Background] Cuthbertson BH, Roughton S, Jenkinson D, Maclennan G, Vale L. Quality of life in the five years after intensive care: a cohort study. Crit Care. 2010;14(1):R6. doi: 10.1186/cc8848. Epub 2010 Jan 20. PMID 20089197
- [Background] Dowdy DW, Eid MP, Dennison CR, Mendez-Tellez PA, Herridge MS, Guallar E, Pronovost PJ, Needham DM. Quality of life after acute respiratory distress syndrome: a meta-analysis. Intensive Care Med. 2006 Aug;32(8):1115-24. doi: 10.1007/s00134-006-0217-3. Epub 2006 Jun 17. PMID 16783553
- [Background] Dowrick AS, Gabbe BJ, Williamson OD, Wolfe R, Cameron PA. A comparison of self-reported and independently observed disability in an orthopedic trauma population. J Trauma. 2006 Dec;61(6):1447-52. doi: 10.1097/01.ta.0000242219.02901.d9. PMID 17159689
- [Background] Gabbe BJ, Cameron PA. Importance of functional and quality of life outcomes in trauma. Surgeon. 2013 Apr;11(2):114. doi: 10.1016/j.surge.2012.11.002. Epub 2012 Nov 27. No abstract available. PMID 23200459
- [Background] Hashem MD, Nallagangula A, Nalamalapu S, Nunna K, Nausran U, Robinson KA, Dinglas VD, Needham DM, Eakin MN. Patient outcomes after critical illness: a systematic review of qualitative studies following hospital discharge. Crit Care. 2016 Oct 26;20(1):345. doi: 10.1186/s13054-016-1516-x. PMID 27782830
- [Background] Herridge MS, Batt J, Hopkins RO. The pathophysiology of long-term neuromuscular and cognitive outcomes following critical illness. Crit Care Clin. 2008 Jan;24(1):179-99, x. doi: 10.1016/j.ccc.2007.11.002. PMID 18241785
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Background] Hodgson CL, Berney S, Harrold M, Saxena M, Bellomo R. Clinical review: early patient mobilization in the ICU. Crit Care. 2013 Feb 28;17(1):207. doi: 10.1186/cc11820. PMID 23672747
- [Background] Hodgson CL, Hayes K, Everard T, Nichol A, Davies AR, Bailey MJ, Tuxen DV, Cooper DJ, Pellegrino V. Long-term quality of life in patients with acute respiratory distress syndrome requiring extracorporeal membrane oxygenation for refractory hypoxaemia. Crit Care. 2012 Oct 19;16(5):R202. doi: 10.1186/cc11811. PMID 23082772
- [Background] Hopkins RO, Herridge MS. Quality of life, emotional abnormalities, and cognitive dysfunction in survivors of acute lung injury/acute respiratory distress syndrome. Clin Chest Med. 2006 Dec;27(4):679-89; abstract x. doi: 10.1016/j.ccm.2006.06.003. PMID 17085255
- [Background] Hopkins RO, Suchyta MR, Farrer TJ, Needham D. Improving post-intensive care unit neuropsychiatric outcomes: understanding cognitive effects of physical activity. Am J Respir Crit Care Med. 2012 Dec 15;186(12):1220-8. doi: 10.1164/rccm.201206-1022CP. Epub 2012 Oct 11. PMID 23065013
- [Background] Innerd P, Catt M, Collerton J, Davies K, Trenell M, Kirkwood TB, Jagger C. A comparison of subjective and objective measures of physical activity from the Newcastle 85+ study. Age Ageing. 2015 Jul;44(4):691-4. doi: 10.1093/ageing/afv062. Epub 2015 May 27. PMID 26018999
- [Background] Iwashyna TJ. Trajectories of recovery and dysfunction after acute illness, with implications for clinical trial design. Am J Respir Crit Care Med. 2012 Aug 15;186(4):302-4. doi: 10.1164/rccm.201206-1138ED. No abstract available. PMID 22896591
- [Background] Kayambu G, Boots R, Paratz J. Physical therapy for the critically ill in the ICU: a systematic review and meta-analysis. Crit Care Med. 2013 Jun;41(6):1543-54. doi: 10.1097/CCM.0b013e31827ca637. PMID 23528802
- [Background] Kulkarni HS, Kulkarni KR, Mallampalli A, Parkar SR, Karnad DR, Guntupalli KK. Comparison of anxiety, depression, and post-traumatic stress symptoms in relatives of ICU patients in an American and an Indian public hospital. Indian J Crit Care Med. 2011 Jul;15(3):147-56. doi: 10.4103/0972-5229.84891. PMID 22013306
- [Background] Lacruz M, Emeny R, Bickel H, Linkohr B, Ladwig Kh. Feasibility, internal consistency and covariates of TICS-m (telephone interview for cognitive status-modified) in a population-based sample: findings from the KORA-Age study. Int J Geriatr Psychiatry. 2013 Sep;28(9):971-8. doi: 10.1002/gps.3916. Epub 2012 Nov 28. PMID 23242951
- [Background] Lea GS, Costello R. Developing an Intensive Care Continuum: incorporating rehabilitation services in critical care. Dimens Crit Care Nurs. 1997 Jan-Feb;16(1):40-6. doi: 10.1097/00003465-199701000-00005. PMID 9016014
- [Background] Lee JJ, Waak K, Grosse-Sundrup M, Xue F, Lee J, Chipman D, Ryan C, Bittner EA, Schmidt U, Eikermann M. Global muscle strength but not grip strength predicts mortality and length of stay in a general population in a surgical intensive care unit. Phys Ther. 2012 Dec;92(12):1546-55. doi: 10.2522/ptj.20110403. Epub 2012 Sep 13. PMID 22976446
- [Background] Luciano JV, Ayuso-Mateos JL, Fernandez A, Serrano-Blanco A, Roca M, Haro JM. Psychometric properties of the twelve item World Health Organization Disability Assessment Schedule II (WHO-DAS II) in Spanish primary care patients with a first major depressive episode. J Affect Disord. 2010 Feb;121(1-2):52-8. doi: 10.1016/j.jad.2009.05.008. Epub 2009 May 22. PMID 19464735
- [Background] Lumb PD. Economic impact of prolonged neuromuscular weakness complicating neuromuscular blockade in the intensive care unit. Crit Care Med. 1996 Oct;24(10):1615-6. doi: 10.1097/00003246-199610000-00002. No abstract available. PMID 8874295
- [Background] Lyons RA, Kendrick D, Towner EM, Christie N, Macey S, Coupland C, Gabbe BJ; UK Burden of Injuries Study Group. Measuring the population burden of injuries--implications for global and national estimates: a multi-centre prospective UK longitudinal study. PLoS Med. 2011 Dec;8(12):e1001140. doi: 10.1371/journal.pmed.1001140. Epub 2011 Dec 6. PMID 22162954
- [Background] Maddox M, Dunn SV, Pretty LE. Psychosocial recovery following ICU: experiences and influences upon discharge to the community. Intensive Crit Care Nurs. 2001 Feb;17(1):6-15. doi: 10.1054/iccn.2000.1536. PMID 11176004
- [Background] McKinley S, Aitken LM, Alison JA, King M, Leslie G, Burmeister E, Elliott D. Sleep and other factors associated with mental health and psychological distress after intensive care for critical illness. Intensive Care Med. 2012 Apr;38(4):627-33. doi: 10.1007/s00134-012-2477-4. Epub 2012 Feb 9. PMID 22318635
- [Background] Myhren H, Toien K, Ekeberg O, Karlsson S, Sandvik L, Stokland O. Patients' memory and psychological distress after ICU stay compared with expectations of the relatives. Intensive Care Med. 2009 Dec;35(12):2078-86. doi: 10.1007/s00134-009-1614-1. Epub 2009 Sep 15. PMID 19756511
- [Background] Needham DM, Davidson J, Cohen H, Hopkins RO, Weinert C, Wunsch H, Zawistowski C, Bemis-Dougherty A, Berney SC, Bienvenu OJ, Brady SL, Brodsky MB, Denehy L, Elliott D, Flatley C, Harabin AL, Jones C, Louis D, Meltzer W, Muldoon SR, Palmer JB, Perme C, Robinson M, Schmidt DM, Scruth E, Spill GR, Storey CP, Render M, Votto J, Harvey MA. Improving long-term outcomes after discharge from intensive care unit: report from a stakeholders' conference. Crit Care Med. 2012 Feb;40(2):502-9. doi: 10.1097/CCM.0b013e318232da75. PMID 21946660
- [Background] Needham DM, Dowdy DW, Mendez-Tellez PA, Herridge MS, Pronovost PJ. Studying outcomes of intensive care unit survivors: measuring exposures and outcomes. Intensive Care Med. 2005 Sep;31(9):1153-60. doi: 10.1007/s00134-005-2656-7. Epub 2005 May 21. PMID 15909169
- [Background] Needham DM, Wang W, Desai SV, Mendez-Tellez PA, Dennison CR, Sevransky J, Shanholtz C, Ciesla N, Spillman K, Pronovost PJ. Intensive care unit exposures for long-term outcomes research: development and description of exposures for 150 patients with acute lung injury. J Crit Care. 2007 Dec;22(4):275-84. doi: 10.1016/j.jcrc.2007.02.001. Epub 2007 Jun 27. PMID 18086397
- [Background] Pandharipande PP, Girard TD, Ely EW. Long-term cognitive impairment after critical illness. N Engl J Med. 2014 Jan 9;370(2):185-6. doi: 10.1056/NEJMc1313886. No abstract available. PMID 24401069
- [Background] Patel RP, Gambrell M, Speroff T, Scott TA, Pun BT, Okahashi J, Strength C, Pandharipande P, Girard TD, Burgess H, Dittus RS, Bernard GR, Ely EW. Delirium and sedation in the intensive care unit: survey of behaviors and attitudes of 1384 healthcare professionals. Crit Care Med. 2009 Mar;37(3):825-32. doi: 10.1097/CCM.0b013e31819b8608. PMID 19237884
- [Background] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324
- [Background] Wasiak J, McMahon M, Danilla S, Spinks A, Cleland H, Gabbe B. Measuring common outcome measures and their concepts using the International Classification of Functioning, Disability and Health (ICF) in adults with burn injury: a systematic review. Burns. 2011 Sep;37(6):913-24. doi: 10.1016/j.burns.2011.02.012. Epub 2011 May 6. PMID 21530087
- [Background] Wilcox ME, Herridge MS. Long-term outcomes in patients surviving acute respiratory distress syndrome. Semin Respir Crit Care Med. 2010 Feb;31(1):55-65. doi: 10.1055/s-0029-1246285. Epub 2010 Jan 25. PMID 20101548
- [Background] Williams TA, Dobb GJ, Finn JC, Knuiman MW, Geelhoed E, Lee KY, Webb SA. Determinants of long-term survival after intensive care. Crit Care Med. 2008 May;36(5):1523-30. doi: 10.1097/CCM.0b013e318170a405. PMID 18434893